CLINICAL TRIAL: NCT02349126
Title: Study of ARC-520 in Patient With Chronic Hepatitis B Virus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to pursue alternative clinical trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Heparc-2005
Record Dates: First submitted 2015-01-20; First posted 2015-01-28 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; HBV infection; Hepatitis B Surface Antigen
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — ARC-520

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): ARC-520 Injection
  Interventions: Drug: ARC-520 Injection

INTERVENTIONS:
Drug: ARC-520 Injection — ARC-520 Injection is a liver-targeted antiviral therapeutic designed to treat chronic hepatitis B virus (HBV) infection via an RNA interference (RNAi) mechanism.
  Other Names: ARC-520

SUMMARY:
Patients with chronic HBV infection will receive ARC-520 in combination with entecavir or tenofovir and be evaluated for safety and efficacy.

DETAILED DESCRIPTION:
This is a single-center, open-label study of ARC-520 in combination with entecavir or tenofovir administered to patients with immune active chronic HBV infection. An iterative trial design is anticipated with potential inclusion of additional cohorts with anticipated enrollment of up to 60 patients. Patients who have signed a Human Research Ethics Committee approved informed consent, and have met all of the protocol eligibility criteria will continue receiving daily oral entecavir (0.5-1.0 mg/day) or daily oral tenofovir (300 mg/day) and a single IV injection of ARC-520. If a serious adverse event (SAE) deemed possibly or probably related to study drug should occur at any point during the study, any further dosing will be put on hold pending a complete review of safety data by the sponsor and the Principal Investigator. Patients will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate, and temperature), weight, AEs, 12-lead ECGs, concomitant medication, blood sample collection for hematology, coagulation, chemistry, PK and exploratory PD measures, HBV virology. Patients will be monitored for a total of 12 weeks. Clinically significant changes including AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the patient is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age
* Written informed consent
* No clinically significant abnormalities at screening/pre-dose 12-lead ECG assessment
* No abnormal finding of clinical relevance
* Diagnosis of immune active chronic HBV infection
* > 6 months of continuous treatment with daily, oral entecavir or tenofovir

Exclusion Criteria:

* Pregnant or lactating
* Acute signs of hepatitis/other infection within 4 weeks of screening
* Antiviral therapy other than entecavir or tenofovir within 3 months of screening
* Prior treatment with interferon or a toll receptor agonist in last 12 months
* Use of anticoagulants, corticosteroids, immunomodulators, or immunosuppressants
* Use of dietary and/or herbal supplements that can interfere with liver metabolism
* Use of any drugs known to induce or inhibit hepatic drug metabolism
* Use of prescription medication or over-the-counter products
* Depot injection/implant of any drug except birth control.
* Known diagnosis of diabetes mellitus.
* History of autoimmune disease
* Human immunodeficiency virus (HIV) infection
* Sero-positive for HCV, and/or history of delta virus hepatitis
* Hypertension: blood pressure > 150/100 mmHg
* History of cardiac rhythm disturbances
* Family history of congenital long QT syndrome/unexplained sudden cardiac death
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease
* History of malignancy, except adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, in situ cervical cancer
* Major surgery within 3 months of screening
* History of alcohol and/or drug abuse < 12 months from screening
* Regularly uses alcohol within past 6 months (ie, more than 14 units of alcohol per week)
* Evidence of acute inflammation, sepsis, or hemolysis
* Diagnosed with a significant psychiatric disorder
* Use of drugs of abuse
* History of allergy to bee venom
* Use of investigational agents/devices within 30 days
* Current participation in an investigational study
* Clinically significant gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease
* History/presence of Gilbert's syndrome, conditions that interfere with absorption, distribution, metabolism, excretion of drugs
* Presence of cholangitis, cholecystitis, cholestasis, or duct obstruction
* Clinically significant history/presence of uncontrolled systemic disease
* Donated blood (500 mL) within 7 days prior to study treatment administration
* History of fever within 2 weeks of screening
* Immunization/planned immunization with live attenuated vaccine except influenza vaccine
* Excessive exercise/physical activity within 7 days of screening/enrolment or during study
* History of coagulopathy or stroke within past 6 months, and/or concurrent anticoagulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy: To evaluate the depth and duration of HBsAg decline in response to a single dose of ARC 520 in combination with entecavir or tenofovir in patients with chronic HBV infection | Through Day 85 post-dosing

SECONDARY OUTCOMES:
Safety:To determine the safety and tolerability of ARC 520 through monitoring of adverse events, vital signs, physical exam changes, blood sampling for hematology, coagulation and chemistry and 12-lead ECGs | Through Day 85 post-dosing
Pharmacokinetic parameters: Cmax, AUC0-24, AUClast, AUCinf, CL, V=CL/kel, kel, t1/2 | Post dosing on Days 1,2 & 3
  Blood samples collected immediately prior to infusion and immediately prior to end of infusion, and 0.5,1,3,6,24,48 hrs post-infusion.
Allergenicity:Evaluate Allergenicity of ARC-520 through Bee Venom Allergy Test (IgE) | Within 30 days prior to first dose and at Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Melbourne, Victoria, Australia